CLINICAL TRIAL: NCT06828003
Title: A Remotely-Delivered Resistance Training Program for Cognitive Function in Men Living With and Beyond Prostate Cancer: A Feasibility Study
Brief Title: Feasibility of a Remotely-Delivered Resistance Training Program for Cognitive Function in Men Living With and Beyond Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Linda Trinh, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 47556
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Resistance Training
Keywords: cancer survivorship; cognitive function; prostate cancer; remote delivery; feasibility; resistance training
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to one of two conditions: resistance training intervention or usual care (i.e., exercise guidelines materials). Participants in the resistance training intervention group will receive a remotely-delivered program two days/week for eight weeks (16 sessions total). One session will be 1:1, led by a qualified exercise professional and completed at home via videoconferencing (i.e., Zoom). The second session will be unsupervised, completed by watching a pre-recorded workout video that will vary bi-weekly to elicit progressive overload and mimic live sessions. Participants randomized to the usual care group will receive exercise guidelines for cancer survivors (i.e., educational materials) from the American College of Sport Medicine via email.
Who Masked: Participant
Masking Description: The participants will only be aware that the researchers are comparing the two conditions, and therefore will be blinded to the study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance Training (Experimental): The resistance training intervention will consist of two remotely-delivered exercise sessions per week for eight weeks (16 sessions total). One session will be a live, remotely delivered 1:1 class led by a qualified exercise professional (~one hour). The second session will be unsupervised, completed by watching a pre-recorded workout video that will vary bi-weekly to elicit progressive overload. Pre-recorded workout videos will be emailed and feature the qualified exercise professional who will provide instruction to mimic live sessions. Both sessions will involve a dynamic warm-up (~10 minutes), 8 resistance-band exercises (~30-45 minutes), followed by a cool-down (~10 minutes).
  Interventions: Behavioral: Resistance Training
- Usual Care (No Intervention): The usual care group will receive exercise guidelines for cancer survivors (i.e., educational material) from the American College of Sport Medicine. Exercise guidelines materials will be provided through email.

INTERVENTIONS:
Behavioral: Resistance Training — The resistance training intervention will consist of two remotely-delivered exercise sessions per week for eight weeks (16 sessions total). One session will be a live, remotely delivered 1:1 class led by a qualified exercise professional (~one hour). The second session will be unsupervised, completed by watching a pre-recorded workout video that will vary bi-weekly to elicit progressive overload. Pre-recorded workout videos will be emailed and feature the qualified exercise professional who will provide instruction to mimic live sessions. Both sessions will involve a dynamic warm-up (~10 minutes), 8 resistance-band exercises (~30-45 minutes), followed by a cool-down (~10 minutes).
  Arms: Resistance Training

SUMMARY:
Prostate cancer and its treatment are associated with many long-term adverse effects including cancer-related cognitive impairment. Specifically, androgen deprivation therapy has been shown to negatively impact cognitive function. Combined aerobic and resistance training has been shown to improve cognitive function in men treated with androgen deprivation therapy, but limited research has observed its impact into survivorship. Additionally, existing study designs are limited to supervised, combined aerobic and resistance training interventions. Remotely-delivered resistance training programs could enhance exercise participation by overcoming commonly reported barriers in men living with and beyond prostate cancer such as transportation, distance to facility, and timing of programs. Alongside the needs to address cancer-related cognitive impairments due to androgen deprivation therapy, resistance training may serve to manage functional deficits, losses in bone mineral density and muscle mass and increases in cardiometabolic risk factors. This study will assess the feasibility of an 8-week remotely-delivered resistance training program to improve cognitive function in men living with and beyond prostate cancer who have a history of androgen deprivation therapy treatment.

DETAILED DESCRIPTION:
Prostate cancer and its treatment are associated with many long-term adverse effects including cognitive impairments which have been shown to improve with combined aerobic and resistance exercise. Existing exercise interventions have reported improved cognitive function for men treated with androgen deprivation therapy (ADT). Many of these studies, however, are limited by subjective measures of cognitive function and the use of a generalized quality of life questionnaire to capture cognitive function. Additionally, existing study designs are limited to supervised, combined aerobic and resistance training (RT) interventions. While combined aerobic and RT interventions elicit improvements in cognitive function following ADT, the independent effects of aerobic exercise and RT is less understood. Alongside the needs to address cancer-related cognitive impairments due to ADT, resistance training may serve to manage functional deficits, losses in bone mineral density and muscle mass and increases in cardiometabolic risk factors. There is indirect evidence to support a role for exercise training to attenuate the negative effects of ADT on cognitive function, however, a lack of research has been conducted with men living with and beyond prostate cancer (LWBPC). Given the unique treatment-related impacts on this patient group, there is a need for more adequately powered randomized controlled trials to investigate the direct effects of exercise, and independent effects of RT, on cognitive function in men LWBPC.

Remotely-delivered interventions may be an effective option to increase exercise among men LWBPC, while enhancing reach and accessibility by overcoming barriers to participation in traditional in-person programs. This includes overcoming some of these commonly reported barriers in men LWBPC including transportation and distance to the facility, the timing of the program, poor weather, and gender- or disease-specific concerns. To address the current gaps in literature, research is needed to assess the feasibility of a remotely-delivered RT program for cognitive function in men living with and beyond prostate cancer. Accordingly, the primary objective of this study is to assess the feasibility (e.g., enrollment, adherence, attrition, safety, participant satisfaction) of an 8-week supervised, remotely-delivered RT program versus usual care (i.e., exercise guidelines materials) for men LWBPC. The secondary objectives of this study are to examine changes in 1) objective cognitive function; 2) subjective cognitive function; 3) physical function; 4) self-reported exercise; and 5) self-reported fatigue. The trial results may be used to inform a larger randomized controlled trial and demonstrate that a remotely-delivered RT program could be an effective supplementary intervention strategy to mitigate the impact of cancer-related cognitive impairment in men LWBPC.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* localized or asymptomatic metastatic primary prostate cancer (i.e., androgen receptor axis agents [ARATs] including conventional ADT, abiraterone, enzalutamide)
* a history of ADT treatment
* not currently undergoing radiation
* no neurological or musculoskeletal co-morbidity inhibiting exercise
* mild cognitive impairment as determined by the TICS-M [scores between 21-24 to separate individuals with mild cognitive impairment and normal cognition (>24)]
* not physically active (self-report <90 minutes of MVPA/week and <2 days of RT/week)
* physician clearance to participate
* access to a webcam and internet
* able to complete the study in English.

Exclusion Criteria:

* a medical condition that prevents unsupervised exercise
* presence of other primary or recurrent invasive cancer
* have experienced a fall in the last 12 months
* use a gait aid device
* current participation in other exercise programs/trials
* colour-blind since the objective cognitive tests require participants to distinguish between colours.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Participant enrollment rate will be one measure of feasibility. Enrollment will be calculated by measuring the number of participants who enrolled in the intervention, divided by the number of participants who were assessed for eligibility
Adherence | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Participant adherence will be one measure of feasibility. Adherence will be measured by assessing the number of exercise sessions attended divided by the total number of exercise sessions that take place (i.e., 16 sessions). Additionally, adherence to the exercise intensity will be reported by assessing the reported RPE and HR of participants during each session.
Attrition | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Attrition will be one measure of feasibility. Attrition will be measured by calculating the number of participants who did not complete the intervention, divided by the number of participants who completed the entirety of the intervention.
Adverse Events | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Adverse events will be one measure of feasibility. This will be assessed as an unexpected and severe medical problem or injury (e.g., cardiac-related events, musculoskeletal injury or pain, falls) that occurs as a result of the intervention.
Participant Satisfaction | Post-intervention (8 weeks).
  A participant satisfaction survey will be administered following the 8-week intervention to assess the acceptability of the intervention by using researcher-generated statements (e.g., "I found the resistance training intervention rewarding"). The survey will assess the burden of the program and the participant's feedback regarding the RT program and overall study experience. Likert scales ranging from 1 (not at all) to 5 (very much) will be used.
Therapeutic Alliance | Post-intervention (8 weeks).
  Therapeutic alliance will be measured using a modified version of the Working Alliance Inventory Short Revised (WAI-SR). Participants will respond to 12-items of statements and questions about experiences participants might have had with their instructor (e.g., [INSTRUCTOR] and I respect each other]. Participants will rate their responses on a scale from 1 (seldom) to 5 (always). Higher scores indicate better therapeutic alliance.

SECONDARY OUTCOMES:
Objective Cognitive Function | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Objective cognitive function will be assessed at baseline and follow-up using the National Institutes of Health (NIH) Toolbox Cognition Battery. The assessment will consist of 5 test instruments: the Picture Sequence Memory Test (episodic memory); the Picture Vocabulary Test (Language-Vocabulary Comprehension); the Oral Reading Recognition Test (Language-Reading Decoding); the List Sorting Working Memory Test (working memory); and the Auditory Verbal Learning Test (working memory). To supplement these tests, the PsyToolkit will be used to deliver the Stroop test (executive function). The cognitive assessments will be delivered remotely via a shared iPad screen and videoconferencing (i.e., Zoom).
Subjective Cognitive Function | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Subjective cognitive function will be assessed at baseline and follow-up using the Functional Assessment of Cancer Therapy-Cognitive Function Version 3 (FACT-Cog v3). This questionnaire will assess cognitive symptoms in the previous 7 days in four domains: perceived impairments, perceived abilities, quality of life, and comments from others. Participants will be asked to rate 37 items related to perceived cognitive complaints on a 5-point Likert scale (0= "not at all" or "never and 4= "very much" or "several times/day) where higher scores indicate fewer cognitive problems and better quality of life.
Physical Function | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Physical function will be measured at baseline and follow-up using the remotely-delivered 30-second sit-to-stand test. The purpose of the 30-second sit-to-stand test is to measure participants' lower body strength and endurance by measuring the number of full chair stands with arms folded at the chest completed in 30-seconds. A qualified exercise professional will oversee timing the participant and counting the number of full stands. Higher scores indicate better physical function.
Self-Reported Exercise | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Self-reported exercise will be measured using the modified Godin Leisure-Time Exercise Questionnaire (GLTEQ). Participants will report the number of times per week and duration that they engage in light, moderate, and vigorous leisure-time exercise, and resistance exercise. Total weekly minutes of MVPA will be calculated as the sum of the number of moderate exercise minutes per week, plus twice the number of vigorous exercise minutes per week. Total RT score will be calculated by summing the number of days spent in RT activities per week.
Self-Reported Fatigue | Change from baseline (pre- intervention) to post-intervention (8 weeks).
  Fatigue will be assessed at baseline and follow-up using the Functional Assessment of Chronic Illness Therapy- Fatigue Scale (FACIT-Fatigue). The FACIT-Fatigue is a 13-item measure will assess self-reported fatigue and its impact upon daily activities and function. Participants will be asked to rate 13 items related to their fatigue in the previous 7 days on a 5-point Likert scale (0="not at all" or "never" and 4= "very much" or "several times/day) where higher scores indicate higher quality of life.
Anxiety and Depression | Baseline (pre- intervention) and post-intervention (8 weeks).
  Anxiety and depression will be assessed at baseline and post-intervention as an exploratory variable using the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item instrument comprised of an anxiety subscale score (HADS-A), a depression subscale score (HADS-D) and a total score (HADS-T), where higher scores indicate higher distress. Each item on the HADS is rated on a 4-point Likert scale, where 0= "not at all" and 3= "yes, definitely".
Clinical Demographics | Baseline (pre-intervention)
  Clinical variables include: cancer type, date of diagnosis, cancer stage, cancer spread, cancer stage, treatment, current treatment status, recurrences, other cancer diagnoses, general health status, comorbidities, concussion history, smoking history, alcohol consumption history.
Age | Baseline (pre-intervention)
  Demographic variable of age will be assessed. Units of measurement is years.
Sex | Baseline (pre-intervention)
  Demographic variable of biological sex will be assessed. Response options are; male and female.
Gender | Baseline (pre-intervention)
  Demographic variable of gender will be assessed. Response options include; agender, bigender/multigender, gender fluid, genderqueer, man, nonbinary, transgender, two-spirit, woman, and other.
Marital Status | Baseline (pre-intervention)
  Demographic variable of marital status will be assessed. Response options are; single, married, common-law, separated, widowed, and divorced.
Highest Level of Education | Baseline (pre-intervention)
  Demographic variable of highest level of education will be assessed. Response options are; some high school, completed high school, some university/college, completed university/college, some graduate school, completed graduate school.
Current Employment Status | Baseline (pre-intervention)
  Demographic variable of current employment status will be assessed. Response options are; disability, retired, part-time, homemaker, full-time, and unemployed.
Ethnicity | Baseline (pre-intervention)
  Demographic variable of ethnicity will be assessed. Response options are; White, Chinese, South Asian, Black or African American, Latin American, South East Asian (Cambodian, Indonesian, Laotian, Vietnamese), Arab, West Asian (Afghan, Iranian), East Asian (Japanese, Taiwan), and other.
Body Mass Index | Baseline (pre-intervention)
  Demographic variable of body mass index will be assessed. Units of measurement are height (ft.) and weight (lb.). Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibeggazene S, Turner R, Rosario D, Bourke L. Remote interventions to improve exercise behaviour in sedentary people living with and beyond cancer: a systematic review and meta-analysis. BMC Cancer. 2021 Mar 24;21(1):308. doi: 10.1186/s12885-021-07989-0. PMID 33761906
- [Background] Dawson JK, Dorff TB, Todd Schroeder E, Lane CJ, Gross ME, Dieli-Conwright CM. Impact of resistance training on body composition and metabolic syndrome variables during androgen deprivation therapy for prostate cancer: a pilot randomized controlled trial. BMC Cancer. 2018 Apr 3;18(1):368. doi: 10.1186/s12885-018-4306-9. PMID 29614993
- [Background] Norris MK, Bell GJ, North S, Courneya KS. Effects of resistance training frequency on physical functioning and quality of life in prostate cancer survivors: a pilot randomized controlled trial. Prostate Cancer Prostatic Dis. 2015 Sep;18(3):281-7. doi: 10.1038/pcan.2015.28. Epub 2015 Jun 16. PMID 26078203
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Amireault S, Godin G, Lacombe J, Sabiston CM. The use of the Godin-Shephard Leisure-Time Physical Activity Questionnaire in oncology research: a systematic review. BMC Med Res Methodol. 2015 Aug 12;15:60. doi: 10.1186/s12874-015-0045-7. PMID 26264621
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Bowman A, Denehy L, Benjemaa A, Crowe J, Bruns E, Hall T, Traill A, Edbrooke L. Feasibility and safety of the 30-second sit-to-stand test delivered via telehealth: An observational study. PM R. 2023 Jan;15(1):31-40. doi: 10.1002/pmrj.12783. Epub 2022 Mar 22. PMID 35138036
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Von Ah D, Tallman EF. Perceived cognitive function in breast cancer survivors: evaluating relationships with objective cognitive performance and other symptoms using the functional assessment of cancer therapy-cognitive function instrument. J Pain Symptom Manage. 2015 Apr;49(4):697-706. doi: 10.1016/j.jpainsymman.2014.08.012. Epub 2014 Sep 18. PMID 25240787
- [Background] Wefel JS, Vardy J, Ahles T, Schagen SB. International Cognition and Cancer Task Force recommendations to harmonise studies of cognitive function in patients with cancer. Lancet Oncol. 2011 Jul;12(7):703-8. doi: 10.1016/S1470-2045(10)70294-1. Epub 2011 Feb 25. PMID 21354373
- [Background] Heaton RK, Akshoomoff N, Tulsky D, Mungas D, Weintraub S, Dikmen S, Beaumont J, Casaletto KB, Conway K, Slotkin J, Gershon R. Reliability and validity of composite scores from the NIH Toolbox Cognition Battery in adults. J Int Neuropsychol Soc. 2014 Jul;20(6):588-98. doi: 10.1017/S1355617714000241. Epub 2014 Jun 24. PMID 24960398
- [Background] Thomas T, Althouse A, Sigler L, Arnold R, Chu E, White DB, Rosenzweig M, Smith K, Smith TJ, Schenker Y. Stronger therapeutic alliance is associated with better quality of life among patients with advanced cancer. Psychooncology. 2021 Jul;30(7):1086-1094. doi: 10.1002/pon.5648. Epub 2021 Mar 8. PMID 33547717
- [Background] Meystre C, Bourquin C, Despland JN, Stiefel F, de Roten Y. Working alliance in communication skills training for oncology clinicians: a controlled trial. Patient Educ Couns. 2013 Feb;90(2):233-8. doi: 10.1016/j.pec.2012.10.013. Epub 2012 Nov 14. PMID 23158787
- [Background] Compen FR, Bisseling EM, Van der Lee ML, Adang EM, Donders AR, Speckens AE. Study protocol of a multicenter randomized controlled trial comparing the effectiveness of group and individual internet-based Mindfulness-Based Cognitive Therapy with treatment as usual in reducing psychological distress in cancer patients: the BeMind study. BMC Psychol. 2015 Aug 13;3(1):27. doi: 10.1186/s40359-015-0084-1. eCollection 2015. PMID 26273472
- [Background] Bar-Sela G, Yochpaz S, Gruber R, Lulav-Grinwald D, Mitnik I, Koren D. The association between the strength of the working alliance and sharing concerns by advanced cancer patients: a pilot study. Support Care Cancer. 2016 Jan;24(1):319-325. doi: 10.1007/s00520-015-2794-6. Epub 2015 Jun 12. PMID 26062924
- [Background] Trinh L, Kramer AF, Rowland K, Strom DA, Wong JN, McAuley E. A pilot feasibility randomized controlled trial adding behavioral counseling to supervised physical activity in prostate cancer survivors: behavior change in prostate cancer survivors trial (BOOST). J Behav Med. 2021 Apr;44(2):172-186. doi: 10.1007/s10865-020-00185-8. Epub 2020 Sep 26. PMID 32979134
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Trinh L, Arbour-Nicitopoulos KP, Sabiston CM, Alibhai SM, Jones JM, Berry SR, Loblaw A, Faulkner GE. A Qualitative Study Exploring the Perceptions of Sedentary Behavior in Prostate Cancer Survivors Receiving Androgen-Deprivation Therapy. Oncol Nurs Forum. 2015 Jul;42(4):398-406. doi: 10.1188/15.ONF.398-406. PMID 26148319
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Colado JC, Garcia-Masso X, Triplett TN, Flandez J, Borreani S, Tella V. Concurrent validation of the OMNI-resistance exercise scale of perceived exertion with Thera-band resistance bands. J Strength Cond Res. 2012 Nov;26(11):3018-24. doi: 10.1519/JSC.0b013e318245c0c9. PMID 22210471
- [Background] Bentvelzen AC, Crawford JD, Theobald A, Maston K, Slavin MJ, Reppermund S, Kang K, Numbers K, Brodaty H, Sachdev P, Kochan NA. Validation and Normative Data for the Modified Telephone Interview for Cognitive Status: The Sydney Memory and Ageing Study. J Am Geriatr Soc. 2019 Oct;67(10):2108-2115. doi: 10.1111/jgs.16033. Epub 2019 Jul 9. PMID 31290146
- [Background] Eng L, Pringle D, Su J, Shen X, Mahler M, Niu C, Charow R, Tiessen K, Lam C, Halytskyy O, Naik H, Hon H, Irwin M, Pat V, Gonos C, Chan C, Villeneuve J, Harland L, Shani RM, Brown MC, Selby P, Howell D, Xu W, Liu G, Alibhai SMH, Jones JM. Patterns, perceptions, and perceived barriers to physical activity in adult cancer survivors. Support Care Cancer. 2018 Nov;26(11):3755-3763. doi: 10.1007/s00520-018-4239-5. Epub 2018 May 29. PMID 29808379
- [Background] Courneya KS, Segal RJ, Gelmon K, Reid RD, Mackey JR, Friedenreich CM, Proulx C, Lane K, Ladha AB, Vallance JK, McKenzie DC. Predictors of supervised exercise adherence during breast cancer chemotherapy. Med Sci Sports Exerc. 2008 Jun;40(6):1180-7. doi: 10.1249/MSS.0b013e318168da45. PMID 18460985
- [Background] Clifford BK, Mizrahi D, Sandler CX, Barry BK, Simar D, Wakefield CE, Goldstein D. Barriers and facilitators of exercise experienced by cancer survivors: a mixed methods systematic review. Support Care Cancer. 2018 Mar;26(3):685-700. doi: 10.1007/s00520-017-3964-5. Epub 2017 Nov 28. PMID 29185105
- [Background] Batalik L, Filakova K, Radkovcova I, Dosbaba F, Winnige P, Vlazna D, Batalikova K, Felsoci M, Stefanakis M, Liska D, Papathanasiou J, Pokorna A, Janikova A, Rutkowski S, Pepera G. Cardio-Oncology Rehabilitation and Telehealth: Rationale for Future Integration in Supportive Care of Cancer Survivors. Front Cardiovasc Med. 2022 Apr 15;9:858334. doi: 10.3389/fcvm.2022.858334. eCollection 2022. PMID 35497988
- [Background] Hojan K, Kwiatkowska-Borowczyk E, Leporowska E, Milecki P. Inflammation, cardiometabolic markers, and functional changes in men with prostate cancer. A randomized controlled trial of a 12-month exercise program. Pol Arch Intern Med. 2017 Jan 10;127(1):25-35. doi: 10.20452/pamw.3888. Epub 2017 Jan 10. PMID 28075422
- [Background] Galvao DA, Taaffe DR, Spry N, Joseph D, Newton RU. Combined resistance and aerobic exercise program reverses muscle loss in men undergoing androgen suppression therapy for prostate cancer without bone metastases: a randomized controlled trial. J Clin Oncol. 2010 Jan 10;28(2):340-7. doi: 10.1200/JCO.2009.23.2488. Epub 2009 Nov 30. PMID 19949016
- [Background] Mundell NL, Daly RM, Macpherson H, Fraser SF. Cognitive decline in prostate cancer patients undergoing ADT: a potential role for exercise training. Endocr Relat Cancer. 2017 Apr;24(4):R145-R155. doi: 10.1530/ERC-16-0493. Epub 2017 Feb 16. PMID 28209634
- [Background] Nguyen PL, Alibhai SM, Basaria S, D'Amico AV, Kantoff PW, Keating NL, Penson DF, Rosario DJ, Tombal B, Smith MR. Adverse effects of androgen deprivation therapy and strategies to mitigate them. Eur Urol. 2015 May;67(5):825-36. doi: 10.1016/j.eururo.2014.07.010. Epub 2014 Aug 2. PMID 25097095
- [Background] Gardner JR, Livingston PM, Fraser SF. Effects of exercise on treatment-related adverse effects for patients with prostate cancer receiving androgen-deprivation therapy: a systematic review. J Clin Oncol. 2014 Feb 1;32(4):335-46. doi: 10.1200/JCO.2013.49.5523. Epub 2013 Dec 16. PMID 24344218
- [Background] Ahmadi H, Daneshmand S. Androgen deprivation therapy for prostate cancer: long-term safety and patient outcomes. Patient Relat Outcome Meas. 2014 Jul 5;5:63-70. doi: 10.2147/PROM.S52788. eCollection 2014. PMID 25045284
- [Background] Trost LW, Serefoglu E, Gokce A, Linder BJ, Sartor AO, Hellstrom WJ. Androgen deprivation therapy impact on quality of life and cardiovascular health, monitoring therapeutic replacement. J Sex Med. 2013 Feb;10 Suppl 1:84-101. doi: 10.1111/jsm.12036. PMID 23387914
- [Background] Ahles TA, Root JC, Ryan EL. Cancer- and cancer treatment-associated cognitive change: an update on the state of the science. J Clin Oncol. 2012 Oct 20;30(30):3675-86. doi: 10.1200/JCO.2012.43.0116. Epub 2012 Sep 24. PMID 23008308